CLINICAL TRIAL: NCT00136968
Title: Assessment of Voriconazole Penetration Into the Brain by Fluorine-Magnetic Resonance Spectroscopy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Mclean Hospital (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A1501060
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Voriconazole

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
The purpose of this study is to determine the amount of voriconazole in the brain by fluorine-magnetic resonance spectroscopy (MRS) and to compare brain levels to plasma levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers 18-55 years of age

Exclusion Criteria:

* Subjects with any condition affecting drug absorption
* Subjects with a positive urine drug screen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-04; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Assess brain levels of voriconazole in the brain using a non-evasive technique of MRS

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer